CLINICAL TRIAL: NCT07288099
Title: Prospective Observational Cohort Study Comparing Recovery Profiles After Target-Controlled Infusion Versus Inhalational Anesthesia in Video-Assisted Thoracoscopic Surgery
Brief Title: Target-Controlled Infusion (TCI) vs Inhalational Anesthesia in Video-Assisted Thoracoscopic Surgery (VATS)
Acronym: TCI-INHALE
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, mert katılmış, Research Assistant, MD, Istanbul University - Cerrahpasa
Other Study IDs: E-24687260-604.01-1455240
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Video-assisted Thoracoscopic Surgery (VATS); Thoracic Surgery, Video Assisted; Postoperative Recovery; General Anesthesia; Anesthesia Techniques
Keywords: Video-Assisted Thoracoscopic Surgery; VATS; Thoracic Surgery; Target-Controlled Infusion; Inhalational Anesthesia; Postoperative Recovery; Extubation Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TCI Group: Patients receiving target-controlled infusion (TCI) anesthesia as part of routine clinical care during VATS procedures. No intervention is assigned by the study team.
- Inhalational Anesthesia Group: Patients receiving inhalational anesthesia (e.g., sevoflurane) as part of routine clinical care during VATS procedures. No intervention is assigned by the study team.

SUMMARY:
This study is designed as a prospective observational cohort to evaluate recovery after video-assisted thoracoscopic surgery (VATS). In our clinic, anesthesia for VATS is commonly provided either with target-controlled infusion (TCI) or with inhalational agents, depending on the routine practice of the anesthesiologist. No randomization or additional intervention will be performed.

During the study period, patients who receive either method as part of standard care will be followed, and perioperative and postoperative data will be recorded. Awakening time, extubation time, Aldrete score progression, pain levels, and early postoperative complications will be compared between the two groups. The aim is to better understand how these widely used anesthesia techniques may influence recovery in VATS patients and to support future clinical decision-making.

DETAILED DESCRIPTION:
This study is planned as a prospective observational cohort carried out in patients undergoing video-assisted thoracoscopic surgery (VATS). In routine practice at our institution, anesthesia for these operations is provided either with target-controlled infusion (TCI)-based total intravenous anesthesia or with inhalational agents. The study will not change the type of anesthesia given to any patient. The method used will depend entirely on the attending anesthesiologist's usual clinical choice.

Patients receiving either technique during the study period will be followed, and perioperative variables will be documented. These include basic demographic data, intraoperative hemodynamic changes, duration of anesthesia, administered drug doses, and oxygenation parameters. Postoperative recovery will be assessed mainly through awakening and extubation times, Aldrete scores, sedation assessments, pain scores, and early complications such as nausea and vomiting.

The purpose of this observational design is to compare the two commonly used anesthesia approaches as they are applied in real clinical practice. By examining postoperative recovery patterns and any differences between groups, the study aims to provide practical information that may help guide anesthesia selection in VATS procedures. No additional risk or intervention will be introduced, and all patient data will be collected in accordance with routine clinical monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years

Patients scheduled for elective video-assisted thoracoscopic surgery (VATS)

ASA physical status I-III

Able to provide informed consent

Planned postoperative recovery in PACU and surgical ward

Exclusion Criteria:

* ASA IV or higher

Hemodynamic or respiratory instability before surgery

Known allergy or contraindication to commonly used anesthetic agents

Neurological or psychiatric conditions that may interfere with recovery assessment

Emergency surgeries

Patients who decline participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing elective video-assisted thoracoscopic surgery (VATS) at our institution. In routine practice, anesthesia for these procedures is provided either with target-controlled infusion (TCI) or with inhalational agents, according to the preference of the attending anesthesiologist. Patients between 18 and 65 years of age who meet the clinical criteria for VATS and are able to give informed consent will be included. Individuals with significant cardiorespiratory instability, ASA IV or higher, or conditions that may interfere with postoperative assessment will not be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Extubation Time | Up to 30 minutes after the end of surgery
  Time from discontinuation of anesthesia to removal of the endotracheal tube. Extubation time will be recorded routinely in the operating room as part of standard postoperative monitoring.

SECONDARY OUTCOMES:
Awakening Time | Up to 20 minutes after surgery
  Time from the end of anesthesia to the patient's first response to verbal command (eye opening or hand squeeze), recorded routinely in the operating room.
Aldrete Score Progression | PACU stay, up to 1 hour
  Aldrete scores will be recorded at standard intervals in the post-anesthesia care unit (PACU) to evaluate early recovery. The time needed to reach an Aldrete score of 9 will be compared between groups.
Postoperative Pain Score (NRS) | First hour after PACU admission
  Numeric Rating Scale (0-10) will be used to assess postoperative pain at PACU admission and during the early postoperative period.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves routinely collected clinical information, and the dataset contains sensitive patient details that cannot be made publicly available. All data will be used only within the study team and stored according to institutional privacy policies.